CLINICAL TRIAL: NCT07376005
Title: Effects of Acute Sugar Intake on Choroidal Thickness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-12-01PS
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Choroid
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral glucose (Active Comparator): Subjects receive 30g of oral glucose
  Interventions: Dietary Supplement: Oral glucose

INTERVENTIONS:
Dietary Supplement: Oral glucose — Participants will consume 30 grams of sugar in the form of glucose tablets.

SUMMARY:
This study aims to bridge that gap by investigating how acute sugar intake influences choroidal thickness.

DETAILED DESCRIPTION:
This investigation will be a prospective, repeated-measures study. All subjects will arrive fasted and will be asked not to consume any outside food or beverages during the three-hour study period, and will be asked to abstain from caffeine intake for 12 hours before participation. A baseline OCT scan of the macula of the right eye will be performed using the Heidelberg Spectralis OCT system. Participants will then consume 30 grams of sugar in the form of glucose tablets. Macular OCT scans of the right eye will be repeated every 30 minutes for 3 hours following sugar consumption.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for enrolment, each subject must have less than 6 diopters of spherical equivalent refractive error, and have no existing diagnosis of diabetes or pre-diabetes.

Exclusion Criteria:

* Any potential subject with known retinal pathology will be excluded. Any potential subject with any other known systemic or ocular conditions that may impact their ability to participate in the study or provide generalizable data will also be excluded.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in choroidal thickness | within 3 hours of baseline
  The primary outcome for this investigation will be changes in choroidal thickness from baseline across timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern College of Optometry, Memphis, Tennessee, United States